CLINICAL TRIAL: NCT05525650
Title: A Randomized, Double Blind, Placebo-controlled, Multiple-dose, Parallel Phase Ⅰ Study to Evaluate Safety and Compare the Immune Stimulating Efficacy of "DF19001" in Dermatophagoides Farinae Sensitized Allergic Rhinitis Volunteers
Brief Title: Comparative Evaluation of Safety and Immune Activity of New Immunotherapeutic Agents for HDM Allergic Rhinitis Patients
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: RAPHAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RapMed 1506-11-A
Record Dates: First submitted 2022-08-16; First posted 2022-09-01 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Mite Allergy; Rhinitis, Allergic; House Dust Mite Rhinitis
Keywords: Microneedle; Micro Array Patch; House Dust Mite Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Antigens, Dermatophagoides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 1Arm A (Experimental): As the maintenance UNIT, 200 PAU
  Interventions: Drug: House Dust Mite Extract, Dermatophagoides Farinae
- 1Arm B (Placebo Comparator): Placebo arm of 1Arm A.
  Interventions: Drug: House Dust Mite Extract, Dermatophagoides Farinae
- 2Arm C (Experimental): As the maintenance UNIT, 400 PAU
  Interventions: Drug: House Dust Mite Extract, Dermatophagoides Farinae
- 2Arm D (Placebo Comparator): Placebo arm of 2Arm C.
  Interventions: Drug: House Dust Mite Extract, Dermatophagoides Farinae
- 3Arm E (Experimental): As the maintenance UNIT, 800 PAU
  Interventions: Drug: House Dust Mite Extract, Dermatophagoides Farinae
- 3Arm F (Placebo Comparator): Placebo arm of 3Arm E.
  Interventions: Drug: House Dust Mite Extract, Dermatophagoides Farinae

INTERVENTIONS:
Drug: House Dust Mite Extract, Dermatophagoides Farinae — [Group 1] Group A receives 100 PAU at week 1 and 200 PAU at week 2 as the induction phase.
  200 PAU is administered for 3 to 16 weeks as a maintenance phase.
  Group B (placebo group) is the placebo arm of group A.
  [Group 2] As the induction phase, group C received 100 PAU at week 1, 200 PAU at week 2, 300 PAU at week 3, and 400 PAU at week 4.
  As the maintenance phase, 400 PAU is administered for 5 to 16 weeks.
  Group D (placebo) is the placebo group in Group C.
  [Group 3] As the induction phase, group E received 100 PAU at week 1, 200 PAU at week 2, 300 PAU at week 3, 400 PAU at week 4, 600 PAU at week 5, and 800 PAU at week 6.
  As the maintenance phase, 800 PAU is administered from 7 to 16 weeks.
  Group F (placebo) is the placebo arm of group E.

SUMMARY:
When administering clinical trial drugs to patients with house dust mite allergic rhinitis, safety/tolerance is comparatively evaluated as the primary outcome, and symptom improvement and immune activity of the disease are comparatively evaluated as secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19 - 65years with allergic rhinitis caused by the house dust mite antigen.
* ImmunoCAP® titer > 3.49 kUA/L for the house dust mite antigen.
* Determined to be suitable for clinical trials as a result of laboratory tests.

Exclusion Criteria:

* Patients with uncontrolled, severe, or moderate asthma according to the Global Initiative for Asthma (GINA) guidelines.
* In case of lactation or pregnancy.
* If an infectious disease that may affect this study is identified.
* Patients with a history of rhinology surgery within 6 months prior to the first administration of the clinical investigational drug.
* If the allergy skin prick test is negative for the house dust mite antigen.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2024-12-21 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Vital signs | 1 day before dosing, Post-study visit(within 15 days after clinical completion)
  Blood pressure (mmHg), Heart rate (BPM), Body temperature(℃)
Health examination | 1 day before dosing, Post-study visit(within 15 days after clinical completion)
  - Physical examination of necessary body parts by interviewing and observing the height (cm), weight (kg), auscultation (lung, heart), and other clinical test subjects
laboratory test | 1 day before dosing, Post-study visit(within 15 days after clinical completion)
  Hematologic examination
laboratory test | 1 day before dosing, Post-study visit(within 15 days after clinical completion)
  Blood coagulation test
laboratory test | 1 day before dosing, Post-study visit(within 15 days after clinical completion)
  Blood chemistry test
Electrocardiography | 1 day before dosing, Post-study visit(within 15 days after clinical completion)
  Measure the 12 lead electrocardiogram. All electrocardiograms are measured after the subject rests for at least 3 minutes in a supine position.
Local Adverse Event | 1 day before dosing, Post-study visit(within 15 days after clinical completion)
  Local adverse events are removed from the subject 4 hours after attaching the clinical trial drug, and the attachment site is photographed and uploaded to the subject's diary (e-diary). The tester evaluates the presence of an adverse reaction through visual evaluation of the photo of the attachment site.
systemic adverse event | 1 day before dosing, Post-study visit(within 15 days after clinical completion)
  Systemic adverse reaction evaluation was evaluated according to the WAO subcutaneous immunotherapy systemic reaction grading system.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No